CLINICAL TRIAL: NCT04559074
Title: Personalised Electronic Record Supported Optimisation When Alone for Patients With Hypertension- Pilot Study for Remote Medical Management of Hypertension During the COVID-19 Pandemic
Brief Title: Personalised Electronic Record Supported Optimisation When Alone for Patients With Hypertension
Acronym: PERSONALCovdBP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Closed Loop Medicine Ltd (Unknown); Innovate UK (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 283209; PERSONAL-Covid BP (Other: Queen Mary University of London); 2020-002494-10 (EudraCT Number); 16393332 (Other: ISRCTN); 283209 (Other: IRAS)
Record Dates: First submitted 2020-08-26; First posted 2020-09-22 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): Intervention group will receive Amlodipine 1mg/ml Oral Solution; starting dose 1-2mg per day for patients not on amlodipine at entry. Participants will take the prescribed dosage daily. Dosage will be reviewed on a fortnightly basis and adjusted as necessary. The total duration is 3 months.
  Interventions: Drug: Amlodipine
- Observational (No Intervention): This group will record blood pressure readings and data on a daily basis for a total of 3 months. They will not take any medication. They will be reviewed on a monthly basis in consultations.

INTERVENTIONS:
Drug: Amlodipine — Amlodipine 1mg/ml Oral Solution; starting dose 1-2mg per day for patients not on amlodipine at entry; starting dose equivalent to current dose for patients on amlodipine at entry or at next 1-2mg dose step (according to clinical need based on the Investigator's judgement). Investigation of whether gradually increasing the dose of liquid amlodipine (can be an add-on to existing amlodipine tablets) in small increments (e.g. 1-2mg) will enable blood pressure control within the sequence 1mg, 2mg, 3mg, 4mg, 5mg, 6mg, 7mg, 8mg, 9mg to a maximum of 10mg amlodipine per day.
  Arms: Interventional

SUMMARY:
This trial is focusing on blood pressure control for patients with high blood pressure (hypertension) during the COVID-19 pandemic when seeing a doctor for advice may be difficult. The study utilises remote consultations by telephone or video conferencing. Patients record blood pressure and data into an electronic diary on their phone which is reviewed in consultations every 2 weeks by a clinician. Medication for this trial is amlodipine as an oral solution which is uptitrated accordingly for patients receiving medication (anticipated 200). 800 patients will be in an observational group recording the same readings and will not receive any medication.

DETAILED DESCRIPTION:
Given the urgent need for effective monitoring and medical management of hypertension during the COVID-19 pandemic, this study will test the feasibility of remote screening and onboarding to remote medical management of hypertension utilizing personalised digital diary record assisted optimisation of Blood Pressure control. Having remote screened a large number of participants, we then test the effect of a very gentle addition of amlodipine 1mg/ml oral solution to the regimes of a subgroup of asymptomatic participants with inadequate BP control.

The majority of participants screened for the study will continue in follow-up and may be offered further developments as may be possible through development of the digital diary and a more comprehensive adaptive protocol which allows for further interventions (such as stop meds at onset of symptoms, or swap on or off ACE/ARB medications etc). Remote monitoring of blood pressure has been shown in times of normal healthcare access to improve blood pressure control, we will assess if the digital diary allows us to help during lockdown/reduced healthcare access and improve blood pressure with amlodipine without the need for blood tests or social contact.

Amlodipine is a calcium-channel blocking drug which reduces blood pressure by relaxing blood vessels (especially veins) but this same effect makes it prone to causing fluid accumulation (oedema) in the lower limbs. There is a large amount of evidence on its effectiveness and safety in reducing blood pressure and in treating stable angina. There appears to be a close relationship between wanted and unwanted effects. Finding the best dose of amlodipine for a patient could be useful in optimizing their blood pressure treatment. At present the tablet doses available are only 5mg and 10mg in the UK. The present study will also investigate the tolerability of side effects and the relationship of these to the prescribed dose of amlodipine. It will measure the side effects of ankle swelling, headache and any other reported side effects using visual analogue scales. The study will utilise a selection of questionnaires to investigate the relationship between participant beliefs about medicines and participants' adherence. The hypothesis of the study is that participants' tolerability of side effects (as measured by VAS) will be related to their beliefs about the necessity of medication (necessity concerns), their concerns about side effects and their adherence to medication.

Participants with uncontrolled blood pressure (systolic =>140 mmHg and/or diastolic =>90 mmHg) on their existing prescription antihypertensive (>= 1 drug) are eligible for the interventional arm of this study. This interventional arm of this study will assess introduction and titration of amlodipine doses within the current maximum licensed dose of 10mg (although higher doses are used in specialist clinics for selected participants). Amlodipine liquid formulation (oral solution) will be used to permit dosing in 1-2mg intervals for optimization of blood pressure control and side effects. Participants will use their standard home blood pressure monitors (a home blood pressure monitor can be provided as appropriate) and will be asked to measure their blood pressure in the morning (three readings) before taking their antihypertensive medication (trough treatment) and again in the evening (three readings).

Participants will participate in remote teleconference consultations (telephone or electronic platform according to participant preference and familiarity, such as Zoom/MS Teams/ WhatsApp/ Facetime) with the William Harvey Clinical Research Centre (WHCRC) at least 2-weekly, following initial (remote) screening with clinical history taking, review of home blood pressure measurements and a thorough review of all information reported by the participant in the digital diary from a 5 day run-in period (see Section 11.6). Remote consultations remain frequent for those participants with poor BP control, but will be less frequent (monthly) for those who have stable blood pressure (defined as above BP<= 140/90) and are followed in the observational arm of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Informed consent.
* Possession of a working smart phone that participant is able to independently use.
* Smartphone to support iOS versions 10.0 and newer or to support Android versions 5.0 (Lollipop) and newer.
* Smartphone to have minimum storage space required to install the digital diary: 250MB.
* Smartphone must have enough memory to run the digital diary.
* Either:
* Participant account of a diagnosis of hypertension consistent with NICE/BIHS criteria on either 24h ABPM or repeated home measures of blood pressure, ideally prior to treatment.

Or •Current treatment with antihypertensive medication.

For the intervention study cohort

* Sub-optimal blood pressure control defined as average systolic blood pressure of 140mmHg or greater, and/or average diastolic blood pressure of 90mmHg or greater during the 5 days run-in period.
* Stable antihypertensive medication during assessment of eligibility.

For the observational study cohort

• Average systolic blood pressure of less than 140mmHg and average diastolic blood pressure of less than 90mmHg during the 5 days run-in period

Exclusion Criteria:

* Current infection, or symptoms suggestive of SARS-2 COVID-19 at the time of screening (rescreening when recovered is allowed).
* Known severe adverse reaction to amlodipine.
* Currently receiving >=10mg /day amlodipine.
* Participation in another clinical trial, where the participant has received IMP in the last three months, with the exception of the MRC Aim-Hy study (IRAS: 199550, REC: 16/EE/0294) where participants can be screened after 6 weeks from final visit.
* Pregnant or lactating or female of childbearing* potential not using adequate contraception (defined as oral contraceptive pill, IntraUterine Device, double barrier methods or abstinence as a clearly defined lifestyle choice).
* Participants who have too limited or no understanding of spoken and/or written English in the opinion of the investigator
* Participants who have hypersensitivity to dihydropyridine derivatives, amlodipine or to any of the excipients.
* Participants with obstruction of the outflow tract of the left ventricle (e.g. high grade aortic grade stenosis).
* Participants with a known intolerance of fructose, sugar, glycerol, maltitol liquid.

(Liquid amlodipine is classed as sugar free, whereas the standard tablet contains lactose).

* Co-morbidities incompatible with study participation e.g. that result in a participant being unable to complete daily entries satisfactorily via his/her smart phone.
* Participants lacking capacity .
* Unstable Heart failure (e.g. after myocardial infarction).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
Reductions in blood pressure in participants with primary hypertension and inadequate BP control by up-titration of amlodipine in 1-2 mg increments. | 3 months
  The primary objective of the study is to assess precision dosing of amlodipine to deliver reductions in blood pressure in participants with primary hypertension and inadequate BP control by up-titration of amlodipine in 1-2 mg increments.

SECONDARY OUTCOMES:
Mean change in daily DBP | 3 months
  Other clinically significant blood pressure measures which related to difference in measured blood pressure between baseline and EOS
Difference between mean changes of blood pressure | 3 months
  Difference between mean changes of blood pressure between interventional and observational cohorts.
Collect data on tolerability / side effects | 3 months
  Reports of side effects using digital diary

CONTACTS AND LOCATIONS:
Overall Officials: David Collier, Principal Investigator — Queen Mary University of London
Locations (2):
- United Kingdom (2):
  - William Harvey Research Institute Clinical Research Centre, Queen Mary University of London, London, London - City of London
  - Queen Mary University London, London

IPD SHARING:
Plan to Share IPD: No
Fully anonymised data will be shared with fellow researchers via conference presentation and via publication of the results in scientific journals. Pseudonymised data will be shared between the research teams named in the application.

REFERENCES:
- [Derived] Collier DJ, Taylor M, Godec T, Shiel J, James R, Chowdury Y, Ebano P, Monk V, Patel M, Pheby J, Pheby R, Foubister A, David C, Saxena M, Richardson L, Siddle J, Timlin G, Goldsmith P, Deeming N, Poulter NR, Gabe R, McManus RJ, Caulfield MJ. Personalized Antihypertensive Treatment Optimization With Smartphone-Enabled Remote Precision Dosing of Amlodipine During the COVID-19 Pandemic (PERSONAL-CovidBP Trial). J Am Heart Assoc. 2024 Feb 20;13(4):e030749. doi: 10.1161/JAHA.123.030749. Epub 2024 Feb 7. PMID 38323513